CLINICAL TRIAL: NCT03045250
Title: Corneal Confocal Microscopy in Patients With Type 1 Diabetes
Acronym: CCM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016-6962
Record Dates: First submitted 2017-01-13; First posted 2017-02-07 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 Diabetes (Active Comparator): Subjects with known Type 1 diabetes
  Interventions: Device: Corneal confocal microscopy; Procedure: Skin biopsy; Procedure: Nerve conduction study; Other: Blood draw
- Healthy Controls (Placebo Comparator): Healthy controls
  Interventions: Device: Corneal confocal microscopy; Procedure: Nerve conduction study; Other: Blood draw

INTERVENTIONS:
Device: Corneal confocal microscopy — Confocal miscroscopy will be used to assess corneal nerve changes due to hyperglycemia.
Procedure: Skin biopsy — Skin biopsy will be used to assess the appearance of nerve fibers in subjects with type 1 diabetes.
  Arms: Type 1 Diabetes
Procedure: Nerve conduction study — Nerve conduction studies will be use to assess for neuropathy.
Other: Blood draw — Subjects will undergo a one time blood draw for biomarkers.

SUMMARY:
Assessing the use of corneal confocal microscopy to evaluate for early neuropathy changes in subjects with Type 1 Diabetes.

DETAILED DESCRIPTION:
Rationale: Poorly controlled diabetes mellitus is associated with microvascular complications, which includes peripheral neuropathy. Peripheral neuropathy associated with diabetes is a painful condition. Its diagnosis is hampered by painful and long nerve conduction studies which fail to diagnose small nerve neuropathy. It is important to study methods of noninvasive methods of early detection, which are sensitive and specific in diagnosing early neuropathy and we propose a novel study that this can be detected in the cornea of the eye.

Aims:

* Estimate corneal small nerve fiber damage in young T1DM subjects (corneal fiber density, nerve branch density, and fiber length) and compare the results to healthy controls using corneal confocal microscopy (CCM).
* Estimate corneal nerve fiber damage in subjects with diabetes, with peripheral neuropathy and subjects with diabetes without peripheral neuropathy, diagnosed by skin biopsies and nerve conduction studies
* Obtain much needed normative values for CCM in adolescents and intraepidermal nerve fiber density from skin biopsies in subjects with type 1 diabetes.
* As a secondary outcome measure, to compare serum biomarkers including leptin, TNF alpha, and fibrinogen in patients with diabetes in those with neuropathy Vs. without neuropathy.

ELIGIBILITY:
Inclusion:

* Subjects with diabetes:
* 18-30 years (cohort 1), adolescents ages 13-17 years (cohort 2).
* Type 1 Diabetes diagnosed via standard ADA criteria

Matched Controls:

* Match for age and gender
* Hemoglobin A1c <6.5%

Exclusion:

For all subjects:

* Contact lens wearers
* Diseases that could damage the cornea, other than diabetes.
* Neurologic disease
* Psychiatric disease
* Amputation
* Foot ulcers
* Pain not of neuropathic origin.
* Presence of Lupus, Sjogren's syndrome and Celiac disease
* Hyperlipidemia requiring lipid-lowering medications
* Peripheral vascular disease
* Neuropathy due to anything besides diabetes
* Presence of any medical condition that may affect nerve conduction (e.g., radiculopathy).

For healthy controls

* Family history of Type 1 Diabetes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Corneal small nerve fiber damage | Assessed one time per subject during study (study completed over 3 years)
  Estimate corneal small nerve fiber damage in young T1DM subjects and compare the results to healthy controls using corneal confocal microscopy (CCM). This will be done by examining the cornea via confocal microscopy and obtaining images. These images will be evaluated looking at how many nerves there are, how they branch, and how long they are).
Normative values for corneal confocal microscopy (CCM) | Assessed one time per subject during study (study completed over 3 years)
  Obtain much needed normative values for CCM in adolescents and intraepidermal nerve fiber density from skin biopsies in subjects with type 1 diabetes. This will be done by obtaining a small biopsy of skin and looking at the number of nerve fibers in the outer layer of the skin.

SECONDARY OUTCOMES:
Serum biomarkers - leptin | Assessed one time per subject during study (study completed over 3 years)
  Measuring serum biomarkers (blood levels) leptin. In participants with diabetes, comparing the blood level measurements of those with neuropathy vs. those without neuropathy.
Serum biomarkers - TNF Alpha | Assessed one time per subject during study (study completed over 3 years)
  Measuring serum biomarkers (blood levels) Tumor Necrosis Factor (TNF) Alpha. In participants with diabetes, comparing the blood level measurements of those with neuropathy vs. those without neuropathy.
Serum biomarkers - fibrinogen | Assessed one time per subject during study (study completed over 3 years)
  Measuring serum biomarkers (blood levels) fibrinogen. In participants with diabetes, comparing the blood level measurements of those with neuropathy vs. those without neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Underland, MD, Principal Investigator — Montefiore Medical Center at Albert Einstein College of Medicine